CLINICAL TRIAL: NCT01834482
Title: A Randomized, Open-label Evaluation of KetoCal® in Initial Combination With the Modified Atkins Diet for the Dietary Management of Intractable Adult Epilepsy.
Brief Title: Modified Atkins Diet Plus KetoCal for Adult Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Nutricia Liverpool (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00068726
Record Dates: First submitted 2013-04-01; First posted 2013-04-18 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Epilepsy; Seizure; Medically Resistant Epilepsy; Medically Resistant Seizures
Keywords: seizures; epilepsy; adult; intractable; medically refractory; Atkins; ketogenic; diet
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Fluid Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Modified Atkins diet plus KetoCal (Active Comparator): Patients will receive the modified Atkins diet in combination with a KetoCal tetrapak daily for the first month. The second month, no tetrapaks will be given.
  Interventions: Dietary Supplement: Modified Atkins diet; Dietary Supplement: KetoCal
- Modified Atkins diet (Active Comparator): Patients will receive the modified Atkins diet for the first month. The second month, they will be given the choice to also use KetoCal in addition to the modified Atkins diet if they choose to do so.
  Interventions: Dietary Supplement: Modified Atkins diet

INTERVENTIONS:
Dietary Supplement: Modified Atkins diet — Patients will receive the modified Atkins diet with a 20 gram per day carbohydrate limit and encouragement to consume plenty of fat and eat to satiety.
Dietary Supplement: KetoCal — Patients will receive a KetoCal 4:1 ratio (fat: carbohydrates and protein) liquid daily for the first month (if randomized to this arm of the study). They will also be started on the modified Atkins diet.
  Other Names: KetoCal 4:1 liquid; KetoCal tetrapak
  Arms: Modified Atkins diet plus KetoCal

SUMMARY:
The modified Atkins diet (MAD) has been shown to be effective in treating children and adults with medically resistant seizures. A recent study in children showed that the use of KetoCal® once per day in addition to the MAD appeared to be beneficial when used during the first month. The investigators hypothesize that including a daily KetoCal® liquid tetrapak with one meal during the initial month of the MAD will produce urinary ketosis in more adult patients than the MAD alone and will lead to greater seizure reduction.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages >17 years.
* At least weekly seizures (or 4 per month). All seizure types allowed.
* Tried at least two anticonvulsants.

Exclusion Criteria:

* Unwilling to restrict carbohydrates
* Significantly underweight (Body Mass Index <18.5)
* Prior use of the modified Atkins diet for ≥ 2 days
* Prior use of KetoCal® at any time for any duration
* Use of the ketogenic diet within the past year
* Kidney disease
* History of hypercholesterolemia (total cholesterol > 300 mg/dl) or hypertriglyceridemia (triglycerides > 200 mg/dl)
* Metabolic or mitochondrial disorder
* Pregnancy or breastfeeding
* Lactose intolerance or milk allergy
* Aversion to liquids or inability to eat solid food

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-03; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Ketosis | 1 month
  Time to urinary ketosis in days will be recorded and whether or not patients achieve serum ketosis at 1 month and 2 months.

SECONDARY OUTCOMES:
Seizure reduction | 2 months
  The percent seizure reduction compared to baseline (1 month before beginning the diet) will be recorded at 1 month and 2 months.
Tolerability and taste | 2 months
  Patients will be asked to rank convenience, taste, texture, and tolerability of the liquid on a 10 point scale (1 = poor, 10 = excellent).
Side effects | 2 months
  Patients will be screened for constipation and asked if they have experienced any side effects related to use of the modified Atkins diet and KetoCal® at 1 and 2 months.
Study completion rate | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Mackenzie C. Cervenka, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Background] Kossoff EH, Dorward JL, Turner Z, Pyzik PL. Prospective study of the modified atkins diet in combination with a ketogenic liquid supplement during the initial month. J Child Neurol. 2011 Feb;26(2):147-51. doi: 10.1177/0883073810375718. Epub 2010 Sep 10. PMID 20833798
- [Background] Cervenka MC, Terao NN, Bosarge JL, Henry BJ, Klees AA, Morrison PF, Kossoff EH. E-mail management of the modified Atkins Diet for adults with epilepsy is feasible and effective. Epilepsia. 2012 Apr;53(4):728-32. doi: 10.1111/j.1528-1167.2012.03406.x. Epub 2012 Feb 14. PMID 22332768
- [Background] Kossoff EH, Rowley H, Sinha SR, Vining EP. A prospective study of the modified Atkins diet for intractable epilepsy in adults. Epilepsia. 2008 Feb;49(2):316-9. doi: 10.1111/j.1528-1167.2007.01256.x. Epub 2007 Oct 5. PMID 17919301
- See also: Adult Epilepsy Diet Center at Hopkins website — http://www.hopkinsmedicine.org/neurology_neurosurgery/specialty_areas/epilepsy/adult/adult-epilepsy-diet-center/